CLINICAL TRIAL: NCT01456780
Title: Relative Efficacy of Loteprednol (Lotemax®) vs. Loteprednol/Tobramycin (Zylet®) in Treatment of Chronic Ocular Surface Inflammation Associated With Meibomian Gland Dysfunction (MGD)/Posterior Blepharitis
Brief Title: Efficacy of Zylet vs. Lotemax for the Treatment of Ocular Surface Inflammation/MGD/Blepharitis
Acronym: ZvL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, Reza Dana, MD, Principal Investigator, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-048H
Record Dates: First submitted 2011-08-02; First posted 2011-10-21 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Meibomian Gland Dysfunction; Posterior Blepharitis
Keywords: Meibomian gland dysfunction; Blepharitis; Dry Eye; Ocular Inflammation; MGD; Zylet; Lotemax; Artificial Tear
MeSH Terms: conditions — Meibomian Gland Dysfunction; Blepharitis; Dry Eye Syndromes | interventions — Loteprednol Etabonate; Tobramycin; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Zylet (Active Comparator): Subject randomized to this arm will be treated with Zylet (Loteprednol/tobramycin), twice a day, for 4 weeks. Zylet is a combination of loteprednol and tobramycin. Loteprednol is in a class of drugs called corticosteroids. Loteprednol inhibits processes in the body that cause inflammation. Tobramycin is an antibiotic.
  Interventions: Drug: Loteprednol/tobramycin
- Lotemax (Active Comparator): Subject randomized to this arm will be treated with Lotemax, twice a day, for 4 weeks. Lotemax is also known as loteprednol. Loteprednol is in a class of drugs called corticosteroids. Loteprednol inhibits processes in the body that cause inflammation.
  Interventions: Drug: Loteprednol
- B+L Advanced Eye Relief Lubricant Drop (Placebo Comparator): Subject randomized to this arm will be treated with B+L Advanced Eye Relief Lubricant Eye Drops (Artificial Tears), twice a day, for 4 weeks.
  Interventions: Drug: B+L Advanced Eye Relief Lubricant Drop

INTERVENTIONS:
Drug: Loteprednol/tobramycin — Zylet (loteprednol/tobramycin) drops, 1 drop twice a day for 4 weeks.
  Other Names: Zylet
  Arms: Zylet
Drug: Loteprednol — Eye drops, 1 drop twice a day for 4 weeks
  Other Names: Lotemax
  Arms: Lotemax
Drug: B+L Advanced Eye Relief Lubricant Drop — Bausch + Lomb (B+L) Advanced Eye Relief Lubricant Drop (Artificial Tears), 1 drop twice a day for 4 weeks.
  Other Names: artificial tears
  Arms: B+L Advanced Eye Relief Lubricant Drop

SUMMARY:
This is a Phase IV, single site, randomized, double masked, parallel control clinical trial of 60 subjects to investigate the variance of efficacy between Lotemax® and Zylet® for treatment of ocular surface inflammation due to meibomian gland dysfunction (MGD). Efficacy will be measured by in-vivo confocal microscopy, corneal fluorescein staining, grading of meibomian gland dysfunction and validated ocular symptom assessment questionnaire.

DETAILED DESCRIPTION:
Posterior blepharitis is a common chronic eyelid condition that is described as generalized inflammation of the posterior lid margin and associated with inflammation of the ocular surface and with symptoms of burning, irritation, and discomfort. Posterior blepharitis is associated with various disorders of the meibomian glands, known collectively as meibomian gland dysfunction (MGD). It is associated either with obstruction and inflammation of the meibomian glands or, less commonly, atrophy of the meibomian glands.

Clinically, MGD often presents with inspissated meibomian glands, oily tear film, as well as inflammation and vascularization of the meibomian gland orifices. Papillary hypertrophy of the tarsal conjunctiva and corneal punctate epitheliopathy are often present, and there are prominent associations with dermatoses, such as acne rosacea, seborrhoeic dermatitis, and atopic dermatitis. Evidence from several sources suggests that MGD of sufficient extent and degree is associated with a deficient tear lipid layer, an increase in tear evaporation, and the occurrence of an evaporative dry eye. In fact MGD is considered to be the most common cause of evaporative dry eye. Individuals with MGD often complain of significant discomfort, including burning, itching, irritation, and photophobia. They may also have other associated symptoms of dry eye and may be plagued by blurred vision, gradual contact lens intolerance. Furthermore, these patients may become functionally handicapped by the negative impact of dry eye on their crucial daily activities such as working, reading, using computer, and driving.

Despite the high incidence of posterior blepharitis, there is currently no consistently effective treatment for this condition and it still remains a therapeutic challenge. Posterior blepharitis has traditionally been managed with eyelid hygiene, topical antibiotics (erythromycin or bacitracin ointments), oral tetracyclines (tetracycline, doxycycline, or minocycline) and corticosteroids which are often time consuming, frustrating, and frequently ineffective or variably effective.

The purpose of this study is to compare the effectiveness of topical loteprednol (corticosteroid) vs. the combination of loteprednol and tobramycin (corticosteroid and antibiotic) against an artificial tear. It is critical to determine to what extent the addition of an antibiotic to a topical steroid can enhance the therapeutic efficacy of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* At least 18 years of age
* Has not worn contact lenses, except for bandage contact lens or rigid gas permeable lens, for at least 2 weeks prior to the study and agrees to not wear contact lenses during study
* Patient is in generally good & stable overall health
* Minimum corneal fluorescein staining of 4 in at least one eye
* OSDI score >22
* The patient must have a diagnosis of posterior blepharitis
* A negative urine pregnancy test result for women of childbearing potential
* Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation.
* Normal lid position and closure
* Ability to understand and provide informed consent to participate in this study
* Willingness to follow study instructions and likely to complete all required visits

Exclusion Criteria:

* History of Stevens-Johnson syndrome or ocular pemphigoid
* History of eyelid surgery
* Intra-ocular surgery or ocular laser surgery within 3 months
* History of microbial keratitis, including herpes
* Active ocular allergies
* Corneal epithelial defect > 1mm2
* Any change in use of topical anti-inflammatories, such as steroids, Restasis, or NSAID within the past 2 weeks
* Any change in dosage of tetracycline compounds (tetracycline, doxycycline, and minocycline) within the past two weeks
* Use of isotretinoin (Accutane) within the past 6 months
* Pregnant or lactating women
* Signs of current infection, including fever and current treatment with antibiotics
* Active liver, renal, or hematologic disease
* The use of any other investigational drug
* Individuals with a known history of glaucoma, individuals with IOP >22 Hg in either eye and individuals with a known family history of glaucoma in primary (first degree) relatives (ie. mother, father, sibling or child)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Dana, MD, MPH, MSc, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye & Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Zylet: Subject randomized to this arm will be treated with Zylet, twice a day, for 4 weeks. Zylet is a combination of loteprednol and tobramycin. Loteprednol is in a class of drugs called corticosteroids. Loteprednol inhibits processes in the body that cause inflammation. Tobramycin is an antibiotic.
  Loteprednol/tobramycin: Zylet (loteprednol/tobramycin) drops, 1 drop twice a day for 4 weeks.
- Bausch & Lomb Lubricant Drops: Subject randomized to this arm will be treated with artificial tears, twice a day, for 4 weeks.
  Bausch + Lomb Advanced Eye Relief Lubricant Eye Drops: Bausch + Lomb Advanced Eye Relief Lubricant Eye Drops (Artificial Tears), 1 drop twice a day for 4 weeks.
Period: Overall Study
Arm/Group | Zylet | Lotemax | Bausch & Lomb Lubricant Drops
Started | 20 | 20 | 20
Completed | 17 | 17 | 20
Not Completed | 3 | 3 | 0
Not completed — Lost to Follow-up | 3 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zylet | Lotemax | Bausch & Lomb Lubricant Drops | Total
Number analyzed (Participants) | 17 | 17 | 20 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (13) | 52 (12) | 57 (12) | 55 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 15 | 32
  Male | 9 | 8 | 5 | 22
Ocular Surface Disease Index [Mean (Standard Deviation); unit: units on a scale] — The Ocular Surface Disease Index score ranges from 0-100, with 100 being severe dry eye symptoms and 0 being no dry eye symptoms
  units on a scale | 59.7 (18.0) | 52.0 (22.6) | 57.0 (21.3) | 56.3 (20.6)
Symptom Assessment in Dry Eye (SANDE) Frequency Score [Mean (Standard Deviation); unit: units on a scale] — The range of the SANDE frequency scale is 0-100, with 0 being the minimum level of frequency of dry eye symptoms and 100 being the maximum level of frequency of dry eye symptoms.
  units on a scale | 77.8 (14.2) | 60.9 (19.4) | 68.1 (17.8) | 68.9 (18.3)
Symptom Assessment in Dry Eye (SANDE) Severity Score [Mean (Standard Deviation); unit: units on a scale] — The range of the SANDE frequency scale is 0-100, with 0 being the minimum level of severity of dry eye symptoms and 100 being the maximum level of severity of dry eye symptoms.
  units on a scale | 67.0 (19.8) | 58.1 (19.6) | 64.2 (19.5) | 63.2 (19.6)
Corneal Fluorescein Staining (CFS) [Mean (Standard Deviation); unit: units on a scale] — The CFS scale ranges from 0 to 15 scale, with 0 representing the minimum level of corneal epitheliopathy and 15 representing the maximum level of corneal epitheliopathy.
  units on a scale | 6.8 (2.6) | 6.6 (2.5) | 6.1 (2.0) | 6.5 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Ocular Surface Disease Index
Description: OSDI is a 12-question survey used to measure the symptoms of dry eye disease. Each of the 12 individual questions rate one symptom on a 0-4 scale, with 4 meaning that the symptom is present all of the time and 0 meaning the symptom is present none of the time. The overall ODSI score is calculated by adding all of the values from the 12 questions, multiplying that value by 25, and dividing the resulting value by the number of questions answered. This results in an overall scale that ranges from 0-100, with 100 being severe dry eye symptoms and 0 being no dry eye symptoms.
Time Frame: Week 4 Time Point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zylet | Lotemax | Bausch & Lomb Lubricant Drops
Number analyzed (Participants) | 17 | 17 | 20
units on a scale | 56.6 (22.4) | 46.4 (24.8) | 48.4 (18.9)

2. Primary Outcome: Symptom Assessment iN Dry Eye (SANDE) Frequency Score
Description: Questionnaire given to patients to assess the frequency of dry eye symptoms. The questionnaire utilizes a 100 mm horizontal Visual Analogue Scale technique to quantify the frequency of the patient's dry eye symptoms. Change is quantified from baseline to week 4. The range of the SANDE frequency scale is 0-100, with 0 being the minimum level of frequency of dry eye symptoms and 100 being the maximum level of frequency of dry eye symptoms.
Time Frame: Week 4 Time Point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zylet | Lotemax | Bausch & Lomb Lubricant Drops
Number analyzed (Participants) | 17 | 17 | 20
units on a scale | 65.9 (28.9) | 51.7 (23.3) | 50.5 (24.3)

3. Primary Outcome: Symptom Assessment iN Dry Eye (SANDE) Severity Score
Description: Questionnaire given to patients to assess the severity of dry eye symptoms. The questionnaire utilizes a 100 mm horizontal Visual Analogue Scale technique to quantify the severity of the patient's dry eye symptoms. Change is quantified from baseline to week 4. The range of the SANDE severity scale is 0-100, with minimum level of severity of dry eye symptoms and 100 being the maximum level of severity of dry eye symptoms.
Time Frame: Week 4 Time Point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zylet | Lotemax | Bausch & Lomb Lubricant Drops
Number analyzed (Participants) | 17 | 17 | 20
units on a scale | 64.5 (25.8) | 54.4 (20.2) | 51.2 (22.0)

4. Primary Outcome: Corneal Fluorescein Staining Score
Description: Corneal Fluorescein Staining is used to assess the level of corneal epitheliopathy that is related to dry eye disease. The CFS scale ranges from 0 to 15 scale, with 0 representing the minimum level of corneal epitheliopathy and 15 representing the maximum level of corneal epitheliopathy.
Time Frame: Week 4 Time Point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zylet | Lotemax | Bausch & Lomb Lubricant Drops
Number analyzed (Participants) | 17 | 17 | 20
units on a scale | 6.3 (4.2) | 5.0 (3.3) | 4.8 (3.2)

ADVERSE EVENTS:
Time Frame: 4 Weeks
Groups:
- Zylet: Subject randomized to this arm will be treated with Zylet, twice a day, for 4 weeks. Zylet is a combination of loteprednol and tobramycin. Loteprednol is in a class of drugs called corticosteroids. Loteprednol inhibits processes in the body that cause inflammation (swelling). Tobramycin is an antibiotic.
  Loteprednol/tobramycin: Zylet (loteprednol/tobramycin) drops, 1 drop twice a day for 4 weeks.
- Lotemax: Subject randomized to this arm will be treated with Lotemax, twice a day, for 4 weeks. Lotemax is also known as loteprednol. Loteprednol is in a class of drugs called corticosteroids. Loteprednol inhibits processes in the body that cause inflammation (swelling).
  Loteprednol: Eye drops, 1 drop twice a day for 4 weeks
Arm/Group | Zylet | Lotemax | Bausch & Lomb Lubricant Drops
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 1/20 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zylet (N=20) | Lotemax (N=20) | Bausch & Lomb Lubricant Drops (N=20)
Eye Pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Blurriness (Eye disorders) | 1 (2) | 1 (1) | 0 (0)
Excess Tearing (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Redness (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Headache (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Shingles (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dryness (Eye disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes